CLINICAL TRIAL: NCT00003216
Title: A Phase III Study of Pre and Post Chemoradiation 5-FU vs. Pre and Post Chemoradiation Gemcitabine for Postoperative Adjuvant Treatment of Resected Pancreatic Adenocarcinoma
Brief Title: Fluorouracil, Gemcitabine, and Radiation Therapy in Treating Patients With Cancer of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-9704; CDR0000066076; E-R9704; SWOG-R9704
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known which treatment regimen is most effective for pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil and gemcitabine plus radiation therapy in treating patients with cancer of the pancreas who have undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall and disease-free survival of patients with resected adenocarcinoma of the pancreas treated with adjuvant fluorouracil-based chemoradiotherapy preceded and followed by fluorouracil vs gemcitabine.
* Compare the local-regional and distant disease control in patients treated with these regimens.
* Compare the acute and late toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to nodal involvement (yes vs no), tumor diameter (less than 3 cm vs 3 cm or greater), and surgical margins (negative vs positive vs unknown). Patients are randomized to one of two treatment arms.

* Arm I: Beginning 3-8 weeks after definitive surgical resection, patients receive fluorouracil IV continuously for 3 weeks. Beginning 1-2 weeks later, patients receive fluorouracil IV continuously concurrently with radiotherapy 5 days a week for 5.5 weeks. Beginning 3-5 weeks after completion of chemoradiotherapy, patients receive fluorouracil IV continuously for 4 weeks every 6 weeks for 2 courses.
* Arm II: Beginning 3-8 weeks after definitive surgical resection, patients receive gemcitabine IV once weekly for 3 weeks. Beginning 1-2 weeks later, patients receive chemoradiotherapy as in arm I. Beginning 3-5 weeks after completion of chemoradiotherapy, patients receive gemcitabine IV once weekly for 3 weeks every 4 weeks for 3 courses.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 518 patients will be accrued for this study within 8.6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Stage T1-4, N0-1 (stage I-IVA)
  * No M1 or NX staging
  * Primary tumor of the pancreas (pancreatic head, neck, uncinate process, or body/tail) and maximum diameter/dimension and tumor status at surgical margin known
* Prior potentially curative gross resection within 3-8 weeks before study
* No non-adenocarcinomas, adenosquamous carcinomas, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct carcinoma, or ampullary carcinoma
* No recurrent disease
* Post-resection CA-19-9 level required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* No significant nausea or vomiting
* No prior malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Able to maintain adequate nutrition (at least 1,500 calories/day)

  * Feeding tube allowed
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 1998-07; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F. Regine, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky; Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center; John S. MacDonald, MD, Study Chair — Beth Israel Comprehensive Cancer Center - West Side Campus
Locations (107):
- United States (106):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Western New York Urology Associates, Buffalo, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Abrams RA, Winter KA, Regine WF, Safran H, Hoffman JP, Lustig R, Konski AA, Benson AB, Macdonald JS, Rich TA, Willett CG. Failure to adhere to protocol specified radiation therapy guidelines was associated with decreased survival in RTOG 9704--a phase III trial of adjuvant chemotherapy and chemoradiotherapy for patients with resected adenocarcinoma of the pancreas. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):809-16. doi: 10.1016/j.ijrobp.2010.11.039. Epub 2011 Feb 1. PMID 21277694
- [Result] Berger AC, Winter K, Hoffman JP, Regine WF, Abrams RA, Safran H, Freedman GM, Benson AB 3rd, Macdonald J, Willett CG. Five year results of US intergroup/RTOG 9704 with postoperative CA 19-9 </=90 U/mL and comparison to the CONKO-001 trial. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):e291-7. doi: 10.1016/j.ijrobp.2012.04.035. Epub 2012 Jun 9. PMID 22682806
- [Result] Farrell JJ, Bae K, Wong J, Guha C, Dicker AP, Elsaleh H. Cytidine deaminase single-nucleotide polymorphism is predictive of toxicity from gemcitabine in patients with pancreatic cancer: RTOG 9704. Pharmacogenomics J. 2012 Oct;12(5):395-403. doi: 10.1038/tpj.2011.22. Epub 2011 May 31. PMID 21625252
- [Result] Regine WF, Winter KA, Abrams R, Safran H, Hoffman JP, Konski A, Benson AB, Macdonald JS, Rich TA, Willett CG. Fluorouracil-based chemoradiation with either gemcitabine or fluorouracil chemotherapy after resection of pancreatic adenocarcinoma: 5-year analysis of the U.S. Intergroup/RTOG 9704 phase III trial. Ann Surg Oncol. 2011 May;18(5):1319-26. doi: 10.1245/s10434-011-1630-6. Epub 2011 Mar 10. PMID 21499862
- [Result] Showalter TN, Winter KA, Berger AC, Regine WF, Abrams RA, Safran H, Hoffman JP, Benson AB, MacDonald JS, Willett CG. The influence of total nodes examined, number of positive nodes, and lymph node ratio on survival after surgical resection and adjuvant chemoradiation for pancreatic cancer: a secondary analysis of RTOG 9704. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1328-35. doi: 10.1016/j.ijrobp.2010.07.1993. Epub 2010 Oct 8. PMID 20934270
- [Result] Tempero MA, Winter KA, Kim GE, et al.: S100A2 as a prognostic marker in patients receiving adjuvant therapy for pancreatic cancer (PC): A secondary analysis of RTOG 9704. [Abstract] J Clin Oncol 29 (Suppl 15): A-4118, 2011.
- [Result] Farrell J, Bae K, Guha C, et al.: Correlation of cytidine deaminase single nucleotide polymorphism and toxicity from gemcitabine in patients with pancreatic cancer from RTOG 9704. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-115, 2009.
- [Result] Farrell JJ, Elsaleh H, Garcia M, Lai R, Ammar A, Regine WF, Abrams R, Benson AB, Macdonald J, Cass CE, Dicker AP, Mackey JR. Human equilibrative nucleoside transporter 1 levels predict response to gemcitabine in patients with pancreatic cancer. Gastroenterology. 2009 Jan;136(1):187-95. doi: 10.1053/j.gastro.2008.09.067. Epub 2008 Oct 7. PMID 18992248
- [Result] Piperdi B, Ng S, Piperdi M, et al.: Single institutional experience with oral capecitabine (Cap) in adjuvant therapy for pancreatic cancer: Gemcitabine (G) followed by Cap/RT followed by G. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-229, 2009.
- [Result] Berger AC, Garcia M Jr, Hoffman JP, Regine WF, Abrams RA, Safran H, Konski A, Benson AB 3rd, MacDonald J, Willett CG. Postresection CA 19-9 predicts overall survival in patients with pancreatic cancer treated with adjuvant chemoradiation: a prospective validation by RTOG 9704. J Clin Oncol. 2008 Dec 20;26(36):5918-22. doi: 10.1200/JCO.2008.18.6288. Epub 2008 Nov 24. PMID 19029412
- [Result] Regine WF, Winter KA, Abrams RA, Safran H, Hoffman JP, Konski A, Benson AB, Macdonald JS, Kudrimoti MR, Fromm ML, Haddock MG, Schaefer P, Willett CG, Rich TA. Fluorouracil vs gemcitabine chemotherapy before and after fluorouracil-based chemoradiation following resection of pancreatic adenocarcinoma: a randomized controlled trial. JAMA. 2008 Mar 5;299(9):1019-26. doi: 10.1001/jama.299.9.1019. PMID 18319412
- [Result] Abrams RA, Winter KA, Regine WF, et al.: Correlation of RTOG 9704 (adjuvant therapy (rx) of pancreatic adenocarcinoma (pan ca)) radiation therapy quality assurance scores (RTQASc) with survival (S). [Abstract] J Clin Oncol 25 (Suppl 18): A-4523, 2007.
- [Result] Berger AC, Winter K, Hoffman J, et al.: Post-resection CA 19-9 predicts overall survival (OS) in patients treated with adjuvant chemoradiation: a secondary endpoint of RTOG 9704. [Abstract] J Clin Oncol 25 (Suppl 18): A-4522, 2007.
- [Result] Regine WF, Garcia M, Berger AC, et al.: Post-resectional CA 19-9 values >90 are associated with significantly worse survival in patients with pancreatic carcinoma treated with adjuvant therapy on RTOG 9704: implications for current and future trials. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-137, S78, 2007.
- [Result] Abrams RA, Winter KA, Regine WF, et al.: RTOG 9704: radiotherapy quality assurance (QA) review and survival. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-39, S22, 2006.
- [Result] Regine WF, Winter KA, Abrams R, et al.: A phase III intergroup trial (RTOG 97-04) of adjuvant pre and post chemoradiation (CRT) 5-FU vs. gemcitabine (G) for resected pancreatic adenocarcinoma. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-42, S23-4, 2006.
- [Result] Regine WF, Winter KW, Abrams R, et al.: RTOG 9704 a phase III study of adjuvant pre and post chemoradiation (CRT) 5-FU vs. gemcitabine (G) for resected pancreatic adenocarcinoma. [Abstract] J Clin Oncol 24 (Suppl 18): A-4007, 180s, 2006.
- [Derived] Reyngold M, Winter KA, Regine WF, Abrams RA, Safran H, Hoffman JP, Mowat RB, Hayes JP, Kessel IL, DiPetrillo T, Narayan S, Chen Y, Ben-Josef E, Delouya G, Suh JH, Meyer J, Haddock MG, Feldman M, Gaur R, Yost K, Peterson RA, Sherr DL, Moughan J, Crane CH. Marital Status and Overall Survival in Patients with Resectable Pancreatic Cancer: Results of an Ancillary Analysis of NRG Oncology/RTOG 9704. Oncologist. 2020 Mar;25(3):e477-e483. doi: 10.1634/theoncologist.2019-0562. Epub 2019 Dec 16. PMID 32162826
- [Derived] Lawrence YR, Moughan J, Magliocco AM, Klimowicz AC, Regine WF, Mowat RB, DiPetrillo TA, Small W Jr, Simko JP, Golan T, Winter KA, Guha C, Crane CH, Dicker AP. Expression of the DNA repair gene MLH1 correlates with survival in patients who have resected pancreatic cancer and have received adjuvant chemoradiation: NRG Oncology RTOG Study 9704. Cancer. 2018 Feb 1;124(3):491-498. doi: 10.1002/cncr.31058. Epub 2017 Oct 20. PMID 29053185